CLINICAL TRIAL: NCT01086215
Title: PEARL II: PEripheral Use of AngioJet® Rheolytic Thrombectomy With a Variety of Catheter Lengths
Brief Title: Registry of AngioJet Use in the Peripheral Vascular System
Acronym: PEARLII
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PEARLII
Record Dates: First submitted 2010-01-20; First posted 2010-03-15 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Peripheral Vascular Disease; Embolism and Thrombosis; Venous Thrombosis
MeSH Terms: conditions — Peripheral Vascular Diseases; Embolism and Thrombosis; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Limb Ischemia: Patients presenting with limb ischemia for treatment
- Deep Vein Thrombosis: Patients presenting with deep vein thrombosis for treatment
- Hemodialysis Access: Patients presenting with thrombosed hemodialysis access for treatment
- Other Thrombotic Conditions: Patients presenting with a thrombotic condition other than limb ischemia, deep vein thrombosis or thrombosed hemodialysis access for treatment

SUMMARY:
The Registry involves the collection of information for research and educational purposes only on the use of AngioJet in the peripheral vascular system.

DETAILED DESCRIPTION:
The PEARL II Registry is a prospective, multi-center, observational registry including 500 patients who meet eligibility from up to 50 sites worldwide. Patient participation will be 12 months including post procedure follow-up contact at 3, 6 and 12 months. The study duration is estimated at 36 months.

A patient's treatment is determined by the treating physician based on the clinical situation and local practices. In contrast to a randomized, controlled trial, there are no pre-defined experimental interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been treated in the peripheral vascular system with any of the AngioJet System catheters.
* Patient has provided appropriate consent/authorization per the site's institutional policy and procedure.

Exclusion Criteria:

* Patient has previously been enrolled in either the PEARL Registry or the PEARL II Registry in the last 12months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community population
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-01; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Blitz, MD, Principal Investigator — Chilton Memorial Hospital; Robert Lookstein, MD, Study Director — Icahn School of Medicine at Mount Sinai; Ali Amin, MD, Principal Investigator — The Reading Hospital & Medical Center
Locations (36):
- United States (32):
  - Phoenix Heart, PLLC, Glendale, Arizona
  - John C. Lincoln Deer Valley Hospital, Phoenix, Arizona
  - Good Samaritan Hospital, Los Angeles, California
  - Christiana Care Health System, Newark, Delaware
  - University of Florida- College of Medicine, Jacksonville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Chris Recknor PC, Gainesville, Georgia
  - Indiana University Health Arnett, Lafayette, Indiana
  - Iowa Health, Des Moines, Iowa
  - Cardiovascular Consultants, Bossier City, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Regional Medical Center of Acadiana, Lafayette, Louisiana
  - Chilton Memorial Hospital, Pompton Plains, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - The University of Toledo Medical Center, Toledo, Ohio
  - St Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - The Reading Hospital & Medical Center, Reading, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - University of South Carolina, Charleston, South Carolina
  - North Central Heart Institute, Sioux Falls, South Dakota
  - Holston Valley Medical Center, Kingsport, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Winchester Medical Center, Winchester, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Winnipeg Regional Health Authority, Winnipeg, Manitoba, Canada
- Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe, Germany
- University of Naples, Naples, Italy
- National Institute of CV Diseases, Bratislava, Slovakia

REFERENCES:
- [Derived] Garcia MJ, Lookstein R, Malhotra R, Amin A, Blitz LR, Leung DA, Simoni EJ, Soukas PA. Endovascular Management of Deep Vein Thrombosis with Rheolytic Thrombectomy: Final Report of the Prospective Multicenter PEARL (Peripheral Use of AngioJet Rheolytic Thrombectomy with a Variety of Catheter Lengths) Registry. J Vasc Interv Radiol. 2015 Jun;26(6):777-85; quiz 786. doi: 10.1016/j.jvir.2015.01.036. Epub 2015 Mar 29. PMID 25824314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting at a participating site who were clinically indicated for a peripheral interventional (arterial, venous or hemodialysis access) procedure with the AngioJet Thrombectomy System were offered the opportuntity to participate. Patients were recruited from January 2010 thru June 2013.
Period: Overall Study
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Started | 212 | 201 | 73 | 14
3 Month Follow Up | 201 (7 LTF; 4 Deaths) | 187 (10 LTF; 4 Deaths) | 64 (5 LTF; 4 Deaths) | 13 (1 LTF; 0 Deaths)
6 Month Follow Up | 192 (5 LTF; 4 Deaths) | 172 (13 LTF; 2 Deaths) | 60 (4 LTF; 0 Deaths) | 12 (1 LTF; 0 Deaths)
12 Month Follow Up | 176 (10 LTF; 6 Deaths) | 154 (16 LTF; 2 Deaths) | 47 (9 LTF; 4 Deaths) | 11 (0 LTF; 1 Death)
Completed | 176 | 154 | 47 | 11
Not Completed | 36 | 47 | 26 | 3
Not completed — Death | 14 | 8 | 8 | 1
Not completed — Lost to Follow-up | 22 | 39 | 18 | 2

BASELINE CHARACTERISTICS:
Population: Descriptive Analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions | Total
Number analyzed (Participants) | 212 | 201 | 73 | 14 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (11.59) | 51.3 (16.37) | 61.6 (13.94) | 56.5 (12.07) | 58.1 (15.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 93 | 36 | 5 | 208
  Male | 138 | 108 | 37 | 9 | 292
Region of Enrollment [Number; unit: participants]
  United States | 154 | 190 | 73 | 13 | 430
  Slovakia | 54 | 11 | 0 | 0 | 65
  Germany | 1 | 0 | 0 | 1 | 2
  Italy | 3 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Degree of Occlusion From Baseline to Final Angiogram/Venogram.
Description: From the Index Procedure's Baseline (pre-endovascular treatment) and Final (post-endovascular treatment) angiograms/venograms, each vessel was assigned a value by the treating physician.
  1. complete occlusion (>90% occlusion);
  2. substantial occlusion (50-90% occlusion OR <50% occlusion and >3cm in length);
  3. partial occlusion (<50% occlusion AND <3cm in length)
  4. patent (without visable thrombus or occlusion) The levels of change (improvement) were calculated by subtracting the baseline assigned angiographic/venographic value from the final value.
Time Frame: Day 1
Population: Intention to Treat (ITT)
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Number analyzed (Participants) | 212 | 201 | 73 | 14
Units on a Scale
  Baseline Value | 1.31 (0.03) | 1.33 (0.03) | 1.36 (0.06) | 1.80 (0.16)
  Final Value | 3.76 (0.04) | 3.73 (0.03) | 3.87 (0.04) | 3.75 (0.12)
  Levels of Change | 2.45 (0.05) | 2.40 (0.04) | 2.50 (0.07) | 1.95 (0.18)
Statistical Analysis 1: Comparison: Limb Ischemia; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Alternative hypothesis is change in occlusion >0
Statistical Analysis 2: Comparison: Deep Vein Thrombosis; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Alternative hypothesis is change in occlusion >0
Statistical Analysis 3: Comparison: Hemodialysis Access; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Alternative hypothesis is change in occlusion >0
Statistical Analysis 4: Comparison: Other Thrombotic Conditions; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Alternative hypothesis is change in occlusion >0

2. Primary Outcome: Rethrombosis
Description: The number of patients affected by rethrombosis of the treated vessels (first episode) throughout a 12 Month Follow-Up.
Time Frame: 3 Month , 6 Month and 12 Month Follow Up
Measure: Number; unit: participants
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Number analyzed (Participants) | 212 | 201 | 73 | 14
participants
  3 Month Follow Up | 21 | 22 | 15 | 0
  6 Month Follow Up | 9 | 4 | 12 | 0
  12 Month Follow Up | 9 | 3 | 7 | 0

3. Secondary Outcome: Concomitant Treatments Used With the AngioJet® System
Description: The # of patients exposed to each treatment option at least once in the given thrombotic condition during the Index Procedure
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Number analyzed (Participants) | 212 | 201 | 73 | 14
participants
  AngioJet Thrombectomy without Lytic | 102 | 94 | 67 | 6
  AngioJet Thrombectomy + Lytic Delivery | 146 | 175 | 15 | 9
  Balloon Angioplasty | 164 | 157 | 69 | 6
  Stent Placement | 124 | 71 | 29 | 2
  Catheter Directed Thrombolysis | 106 | 143 | 0 | 2
  Atherectomy | 9 | 0 | 0 | 0
  Filter Placement | 17 | 51 | 0 | 0
  Non AngioJet Thrombectomy | 31 | 14 | 45 | 2

ADVERSE EVENTS:
Time Frame: Index Procedure thru 12 Month Follow Up
Description: Events that were related to the initial Index Procedure and/or AngioJet
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Serious Adverse Events (participants affected / at risk) | 2/212 | 2/201 | 0/73 | 0/14
Other Adverse Events (participants affected / at risk) | 0/212 | 0/201 | 0/73 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Limb Ischemia (N=212) | Deep Vein Thrombosis (N=201) | Hemodialysis Access (N=73) | Other Thrombotic Conditions (N=14)
Bleeding Requiring Transfusion (Surgical and medical procedures) | 2 | 1 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less